CLINICAL TRIAL: NCT01366001
Title: A Phase 1, Multiple-dose, Parallel Group Study to Evaluate the Safety and Pharmacodynamic Effects of RDC-0313-buprenorphine (ALKS 33-BUP) Administered Alone and Co-administered With Cocaine to Opioid-experienced Cocaine Abusers
Brief Title: ALK33BUP-101: Safety and Pharmacodynamic Effects of ALKS 33-BUP Administered Alone and When Co-administered With Cocaine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: ALK33BUP-101; R01DA031000 (NIH)
Record Dates: First submitted 2011-06-02; First posted 2011-06-03 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Cocaine Abuse
Keywords: Opioid; Cocaine; Dependence; Abuse; Intravenous; Buprenorphine
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ALKS 33-BUP (Experimental)
  Interventions: Drug: ALKS 33-BUP
- ALKS 33 (Experimental)
  Interventions: Drug: ALKS 33
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALKS 33-BUP — Sublingual administration, ALKS 33 + buprenorphine, administered once daily for 10 consecutive days.
  Other Names: ALKS 33-BUP: RDC-0313 + buprenorphine.
  Arms: ALKS 33-BUP
Drug: ALKS 33 — Sublingual administration, ALKS 33 administered once daily for 10 consecutive days.
  Other Names: ALKS 33: RDC-0313.
  Arms: ALKS 33
Drug: Placebo — Sublingual administration, Placebo administered once daily for 10 consecutive days.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of ALKS33-BUP when administered to opioid-experienced cocaine abusers.

DETAILED DESCRIPTION:
There are no currently available pharmacologic treatments for cocaine abuse and/or dependence and the unmet medical need is growing. In collaboration with the National Institute on Drug Abuse (NIDA), Alkermes, Inc. is investigating a fixed-dose combination product consisting of ALKS 33 (also referred to as RDC-0313) and buprenorphine (ALKS 33-BUP) for the treatment of cocaine abuse and/or dependence (Grant Number R01DA031000).

This is a randomized, double-blind, placebo-controlled, parallel design inpatient study. Eligibility will be established which includes responses to cocaine infusions at baseline, prior to study drug administration. Approximately 30 opioid-experienced cocaine abusers will be randomized 1:1:1 to receive study drug. Study drug will be administered once daily for 10 consecutive days. Pharmacodynamic assessments and drug-drug interactions will be closely monitored during the study. Following study drug administration, subjects will receive cocaine infusions to evaluate the effect of treatment on the subjective effects and the PK/PD of cocaine. Subjects will be discharged from the clinical research unit 2 days after the last infusion of cocaine. Subjects will return for follow-up between 7 and 14 days after discharge. The full study will take subjects approximately 28 days, with 17 days of inpatient stay.

ELIGIBILITY:
Inclusion Criteria

In order to participate in the study, subjects must:

1. Be volunteers who are not seeking treatment for drug addiction.
2. Be between 21 and 50 years of age, inclusive.
3. Have a body mass index (BMI) within the range of 18.0 to 30.0 kilograms per square meter (kg/m2), inclusive, and a minimum weight of at least 50.0 kilograms(kg) at screening.
4. Have experience using cocaine by the smoked or IV route within the past year, and a positive urinary drug screen for cocaine prior to study intake.
5. Have opioid experience within 3 years, and not physically dependent on opioids as confirmed by a naloxone challenge.
6. Be able to verbalize understanding of the consent form, able to provide written informed consent, and verbalize willingness to complete study procedures, prior to the initiation of any protocol-specific procedures.
7. Have a medical history and physical examination that demonstrate no clinically significant contraindication for participating in the study.
8. Pass qualification criteria for response to IV cocaine infusions.

Exclusion Criteria

In order to participate in the study, subjects must not:

1. Have a current or past history of seizure disorder, including alcohol- or stimulant-related seizure, febrile seizure, or significant family history of idiopathic seizure disorder. Have any previous clinically significant reaction to cocaine, including loss of consciousness or seizure.
2. Other than drug abuse, have any history of clinically significant major psychiatric illness (eg, severe mood disorder, psychotic disorders ) according to the Diagnostic and Statistical Manual, Fourth Edition, Text Revision(DSM IV-TR)criteria or disorders secondary to drug use in the opinion of the investigator.
3. Present with symptoms of withdrawal following administration of the naloxone challenge test.
4. Have a history of liver disease or current elevation of aspartate aminotransferase (AST) or alanine aminotransferase (ALT) exceeding 3x the upper limit of normal.
5. Have a history of allergy or hypersensitivity to opioid agonists (eg, buprenorphine) or opioid antagonists (eg, naltrexone, naloxone).
6. Have a history of hepatitis C, or human immunodeficiency virus (HIV) types 1 and/or 2.
7. Have a positive urine drug screen upon screening for drugs other than cocaine (or bioequivalent metabolite), marijuana (tetrahydrocannabinol, THC), or due to their long-elimination half-life, benzodiazepines.
8. Have a positive alcohol test at screening or at admission to the inpatient phase of the study. If a subject presents with positive alcohol test, the subject can be rescheduled at the discretion of the sponsor and the investigator or designee.
9. If female, be currently pregnant or lactating or planning to become pregnant within 60 days of last study drug administration.
10. Have any clinically significant history of cardiac disease, including cardiovascular and conduction abnormalities or electrocardiogram (ECG) evidence of cardiac abnormalities.
11. Have used cocaine exclusively through the intranasal route.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2011-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
The primary outcome measures are safety and pharmacokinetics (PK)/ pharmacodynamics (PD) | Study drug will be administered once daily for 10 consecutive days.
  For safety, the primary outcome measures are AEs and cardiovascular responses (Heart Rate, Blood Pressure, Electrocardiogram) collected during cocaine infusions at baseline and during treatment with ALKS 33-BUP, ALKS 33 and placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard L. Silverman, MD, Study Director — Alkermes, Inc.
Locations (1):
- Alkermes Study Site, Overland Park, Kansas, United States